CLINICAL TRIAL: NCT03591653
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of LXI-15028 in the Treatment of Non-erosive Reflux Disease in Chinese Patients for 4 Weeks
Brief Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo Controlled Phase III Study to Evaluate the Efficacy and Safety of LXI-15028 in Non-erosive Reflux Disease in Chinese Patients for 4 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC821603
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LXI-15028 50mg group (Experimental)
  Interventions: Drug: LXI-15028
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LXI-15028 — The investigational products are administrated orally, once in the morning every day, and each dose includes one tablet of investigational products (LXI-15028 50mg active agent or placebo). If the investigational product is not taken in the morning, subjects can take it before 6:00 p.m. on the same day. The duration of treatment is 4 weeks.
  Arms: LXI-15028 50mg group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This is one multi-center, randomized, double-blind, parallel-group, placebo controlled Phase III clinical study to evaluate the efficacy and safety of LXI-15028 50 mg in treatment of non-erosive reflux disease in Chinese patients for 4 weeks.

Screening-eligible subjects will be randomized into LXI-15028 50mg group or placebo group at Visit 2 (Day 0) according to the ratio of 1:1 and receive study treatment for 4 weeks. They will start to take the investigational products in the following morning of Visit 2 (Day 1) and start to complete the subject's diary from the day of study treatment initiation. After 2 weeks of study treatment, subjects will return to the study site and complete Visit 3, after which receive study treatment for another 2 weeks and then complete Visit 4. On the day of Visit 4, subjects will not take any drug. All the subjects will be followed up by phone (Visit 5) at Day 28±3 after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Subject who volunteers to sign the written informed consent form approved by the independent ethics committee and agrees to participate in this study prior to the initiation of any study procedures.
* Subject who is able to understand and follow the protocol requirements and agrees to participate in all the study visits.
* Male or female subjects with age ≥ 18 years.
* Having experienced heartburn (burning or pain behind the breastbone) and regurgitation (acid taste in the mouth and discomfort movement of materials upwards from the stomach) symptoms at least three months prior to screening.
* Having experienced heartburn and regurgitation within 7 days prior to screening, with the frequency and severity in symptom assessment meeting at least one of the following items:

  * Mild heartburn for at least 2 days, with regurgitation;
  * Mild regurgitation for at least 2 days, with heartburn;
  * Moderate or more severe heartburn for at least 1 day, with regurgitation;
  * Moderate or more severe regurgitation for at least 1 day, with heartburn. (Note: To be determined by using the RDQ [item a, b, e, f] completed by subject.) And the RDQ symptom assessment before randomization (Visit 2) still meets the above criteria.
* Within 14 days before study initiation, the subject has been confirmed with no mucosal damage through upper gastrointestinal endoscopy based on Los Angeles (LA) classification. And non-erosive reflux disease is clinically diagnosed by the investigator.
* Subject who agrees to use appropriate medical method for contraception from the signature of the informed consent form to 28 days after the last dose of study medication (not including women in medically sterile state):

  * Women under medically sterile state can participate in this study, for example, postmenopausal state (spontaneous amenorrhea at least for 12 months), post hysterectomy, post bilateral salpingectomy and post bilateral oophorectomy;
  * Appropriate medical contraceptive measures include intrauterine device, physical barrier (male condom, female condom), subcutaneous implant, sustained release contraceptive injection, bilateral salpingectomy and bilateral vasoligation. Note: Use of oral contraceptives is not allowed during the course of study, and dual contraceptive methods are recommended, as to ensure no occurrence of pregnancy during the course of study.

Exclusion Criteria:

* Subject who had participated in this study previously, or had participated in other P-CAB drug clinical studies.
* Participation in other clinical study within 3 months prior to screening, except for the two following circumstances:

  * The study which the subject is participating or participated in is a non-interventional study (e.g. observational study or questionnaire survey) and is judged by investigators to have no interference with the efficacy and safety evaluation in the present study;
  * Subject had signed the informed consent form and participated in another study (NC821602) sponsored by this sponsor in the same study site, but had been withdrawn from that study prior to the start of any treatment.
* Subjects who participate in the plan or conduction of this study (e.g., the sponsor or staff of the study site).
* Women who are pregnant or lactating.
* Subject who is known to be allergic to the active ingredient or Talcid® of the investigational product (including esomeprazole).
* Subject who is unable to undertake an upper gastrointestinal endoscopy.
* Subject who is unable to complete the subject's diary by oneself.
* Subject who has history of manic-depression, anxiety disorder, panic disorder, somatoform disorder, personality disorder or other mental disorder.
* Subject who is diagnosed as erosive esophagitis, acute upper gastrointestinal bleeding, gastric ulcer or duodenal ulcer within two months prior to screening.
* Subject who has symptoms such as odynophagia, serious dysphagia, bleeding, decreased body weight, anemia or hematochezia that represent "warning" to presume gastrointestinal malignant disease, unless the possibility of the malignant disease is excluded through an endoscopy.
* History of malignant tumor within 5 years prior to screening (if the subject's basal cell carcinoma or cervical carcinoma in situ has been cured, he/she will be allowed to participate in this study).
* Subject who is diagnosed as achalasia of the cardia, secondary esophageal motility disorder, irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), Zollinger-Ellison syndrome or eosinophilic esophagitis.
* Subject with history of gastrointestinal surgery, except simple fenestration, appendectomy, cholecystectomy or endoscopic resection of benign tumor.
* Subject who plans to be hospitalized for receiving selective surgery during the study.
* Subject with non-reflux-related esophageal stenosis, hiatus hernia, gastroesophageal varices, active peptic ulcer, gastric bleeding or malignant tumor that is found in upper gastrointestinal endoscopy.
* Subject with uncontrolled and unstable hepatic, renal, cardiovascular, respiratory, endocrine or central nervous system disease as judged by investigators.
* Subject with history of chronic alcohol consumption (more than 14 cups per week, each cup corresponds to 360 mL beer or 150 mL wine or 45 mL liquor) or drug abuse within 5 years prior to screening.
* Use of any PPI, P-CAB or other drugs related to the treatment of GERD (including H2-receptor antagonist, prostaglandin or mucosal protective agent), or any other antiemetic, emetic drugs within two weeks prior to the initiation of study treatment.
* Subject who needs non-steroidal anti-inflammatory drugs (NSAIDs) during the study, unless the subject had started to use low dose aspirin (≤ 100 mg/day) prior to screening.
* Use of potent-to-moderate cytochrome metabolism enzyme CYP3A4 inhibitor or inducer within 4 weeks prior to study treatment, including but not limited to the following drugs:

  * CYP3A4 inhibitors: Ketoconazole, Indinavir, Saquinovir, Atazanavir, Amprenavir, Fosamprenavir, Nefazodone, Itraconazole, Telithromycin, Fluconazole, Troleandomycin, Cimetidine, Aprepitant, Fluvoxamine, Amiodarone, Ritonavir, Erythromycin, Clarithromycin, and Diltiazem;
  * CYP3A4 inducers: Barbiturate, Phenytoin, Rifampin, St John's wort, Carbamazepine, Dexamethasone, Rifabutin, and Phenobarbital etc.
* Subject currently using antipsychotic drug, antidepressant agent or anti-anxiety agent.
* Any of the following laboratory abnormalities at screening:

  * AST≥2 x upper limit of normal (ULN);
  * ALT≥2 x ULN;
  * ALP≥2 x ULN;
  * γ-GT≥2 x ULN;
  * Total bilirubin ≥2 x ULN;
  * BUN (or urea) ≥1.5 x ULN;
  * Creatinine ≥1.5 x ULN.
* Subject with clinically significant abnormality in ECG at screening, including serious arrhythmia, multifocal premature ventricular contraction (PVC), second degree or above atrioventricular block, prolonged QT interval (QTc ≥ 450 ms for male, QTc ≥ 470 ms for female).
* Current infection of human immune deficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) confirmed by tests.
* Judged by the investigator, there are other conditions rendering the subject's illegibility for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Resolution of main symptoms | 4 weeks after receiving oral doses
  Resolution rate of main symptoms (heartburn, regurgitation) at Week 4: percentage of patients with complete resolution of main symptoms (for consecutive 7 days) at Week 4. Note: At Week 4, Reflux Disease Questionnaire (RDQ) (item a, b, e, f) is used to evaluate all main symptoms during previous consecutive 7 days. Complete resolution is defined as the main symptoms are completely resolved and do not occur.

SECONDARY OUTCOMES:
Resolution of main symptoms | 2 week after receiving oral doses
  Resolution rate of main symptoms (heartburn, regurgitation) at Week 2: percentage of patients with complete resolution of main symptoms (for consecutive 7 days) at Week 2. The main symptoms are evaluated using RDQ.
Symptom improvement | 4 weeks after receiving oral doses
  Change of Reflux Disease Questionnaire (RDQ) score (including severity score and frequency score) of each post-treatment visit from baseline;Symptom assessment based on subject diary;
Life quality improvement | 4 weeks after receiving oral doses
  Change of Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) score of each post-treatment visit from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Doctor, Principal Investigator — Changhai Hospital Shanghai
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided